CLINICAL TRIAL: NCT03655535
Title: Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Effect of BTI320 in Addition to Current Treatment With Metformin and/or Sulfonylureas on Glycemic Control in Subjects With Type 2 Diabetes
Brief Title: Multicenter Study to Evaluate the Effect of BTI320 on Glycemic Control in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Therapeutics (Industry)
Collaborators: Sugardown Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTI320-SG02
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Type2 Diabetes Mellitus
Keywords: BTI320; Sugardown; Post-prandial glucose excursions
MeSH Terms: interventions — PAZ320

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: randomized, placebo-controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BTI320 (Experimental): 4 g BTI320 administered 10 min before breakfast, lunch, and dinner
  Interventions: Drug: BTI320
- Placebo (Placebo Comparator): Placebo administered 10 min before breakfast, lunch, and dinner
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BTI320 — Non-systemic galactomannan complex polysaccharide
  Other Names: Sugardown; PAZ320
  Arms: BTI320
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of the current study is to investigate the efficacy and safety of BTI320 compared to placebo in addition to metformin and/or sulfonylureas on glycemic control over 12 weeks in subjects with type 2 diabetes mellitus. This is a randomized, placebo-controlled, double-blind, multi-center study with two treatment arms. Study duration will be approximately 12 weeks. Participants will ingest 4 g BTI320 or matching placebo approximately 10 minutes before starting a meal, 3 times per day, at breakfast, lunch, and dinner. Eight study visits will be scheduled after the Screening visit: Baseline (day 0), weeks 3, 6, and 12 (Visits 2, 4, 6, and 8 respectively) for safety and efficacy assessments and Visits 3, 5, 7 and 9 to remove the Continuous Glucose Monitoring System.

DETAILED DESCRIPTION:
The objective of the current study is to investigate the efficacy and safety of BTI320 compared to placebo in addition to metformin and/or sulfonylureas on glycemic control over 12 weeks in subjects with type 2 diabetes mellitus. This is a randomized, placebo-controlled, double-blind, multi-center study with two treatment arms. Study duration will be approximately 12 weeks. Participants will ingest 4 g BTI320 or matching placebo approximately 10 minutes before starting a meal, 3 times per day, at breakfast, lunch, and dinner. Participants will be instructed not to take the Investigational Medicinal Product with other drugs at the same time. Additional mealtime medication must be taken after consumption of the meal. A nutritionist, dietitian, or study personnel will provide instructions to subjects regarding dietary intake and the need to keep a detailed food record in an online calorie counter and have it entered into an electronic data capture during the study period. In general, subjects will be asked to follow normal meal plans recommended to patients with diabetes. Non-compliance will be defined as taking <80% or >120% of Investigational Medicinal Product during any outpatient evaluation period (visit to visit). Subjects who are non-compliant will be replaced to meet the goal of 60 evaluable subjects. Eight study visits will be scheduled after the Screening visit: Baseline (day 0), weeks 3, 6, and 12 (Visits 2, 4, 6, and 8 respectively) for safety and efficacy assessments and Visits 3, 5, 7 and 9 to remove the Continuous Glucose Monitoring System.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old.
* Established type 2 diabetes as assessed by:

  * Fasting blood glucose (>126 mg/dL/7 mmol/L), or
  * 2 hr oral glucose tolerance test (>200 mg/dL/11.1 mmol/L), or
  * HbA1c is ≥7.0% within 3 months of enrollment and on a stable dose of metformin and/or sulfonylureas for at least 12 weeks.
* Body Mass Index (BMI) >23 kg/m2.
* Treated with metformin and/or sulfonylureas (monotherapy or combination therapy) stable and maximally tolerated for at least three months prior to study participation. Subjects should be on stable and maximally tolerated doses throughout the study unless sulfonylureas require adjustment to reduce the risk of hypoglycemia during the study.
* Subjects who are otherwise in generally satisfactory health.
* Likely to follow study requirements, in particular, to adhere to maintaining a suitable diet and keeping an online diary of their food intake and weight measured once weekly via EDC.
* Female subjects have negative urine pregnancy test at the Screening visit.
* Provides signed informed consent to participate in the study. Informed consent must be given by the subject prior to inclusion in the study, and before performing any study procedures, including the screening visit.

Exclusion Criteria:

* Have type 1 diabetes (insulin-dependent diabetes mellitus [IDDM]).
* Treated with long-acting glucagon-like peptide-1 (GLP-1) receptor agonists, dipeptidyl peptidase-4 (DPP-4) inhibitors, alpha-glucosidase inhibitor, regular insulin, rapid-acting insulin analog, or sodium-glucose cotransport-2 inhibitors (SGLT-2). Treatment with any of these drugs should have been stopped at least 3 months before inclusion.
* Current or recent (within past 30 days) participation in another investigational drug or device study.
* Have participated in a previous study of BTI320.
* Have any uncontrolled cardiovascular risk factors (hypertension, hyperlipidemia), past clinical manifestation of coronary artery disease, blood dyscrasias, or significant cerebrovascular disease in the previous year. Any concomitant drug treatment for a condition not related to diabetes should be discussed and approved with the study Medical Monitor.
* Pregnant or breastfeeding, or plan to become pregnant within one year after randomization.
* Food allergy or severe food intolerance assessed by the Principal Investigator.
* History of allergy or intolerance to BTI320 (PAZ320 or SugarDown) or equivalent.
* Have known condition(s) influencing their glycemic levels (e.g. Cushing syndrome, pancreatic diseases, acromegaly).
* Have human immunodeficiency virus (HIV) infection, hepatitis, tuberculosis, or other serious infectious disease.
* History of alcohol addiction or drug abuse (illegal or controlled pharmaceutical substances) within past year prior to randomization.
* Have planned major surgery within 6 months after randomization.
* Have a terminal illness.
* Serum creatinine of >1.4 mg/dL (>124 μmol/L) in women or >1.5 mg/dL (>133 μmol/L) in men or subjects with end-stage renal disease (Estimated Glomerular Filtration Rate calculated by CKD-EPI [eGFR] <10 mL/min/1.73 m2).
* Have serum Alanine Aminotransferase (SGPT) >3 times upper limit of normal.
* History of cancer, other than non-melanoma skin cancer, that requires treatment during the previous five years prior to randomization.
* History of hemolytic anemia, repeated blood transfusions, or other conditions making HbA1c results unreliable as an indicator of chronic glucose level; hematocrit (Hct) <35% for men and <33% for women.
* History of solid organ transplant.
* Treatment with systemic glucocorticoids (except for short-term therapy [5 days or less]).
* Treatment with atypical anti-psychotics.
* In the opinion of the principal investigator, the subject is unlikely to follow the study protocol.
* Employment/lifestyle that requires nocturnal hours.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
2 hr PPG | Week 12
  Change from baseline to week 12 in area under the curve (AUC) 2-hr post-prandial glucose (PPG) excursions in subjects receiving BTI320 compared with those subjects receiving placebo.

SECONDARY OUTCOMES:
HbA1c | Weeks 3, 6, and 12
  Change in Hemoglobin A1c (HbA1c) serum levels from baseline
2 hr PPG | Weeks 3 and 6
  Change from baseline of AUC 2-hr PPG
1 hr PPG | Weeks 3, 6, and 12
  Change from baseline of AUC 1-hr PPG
3 hr PPG | Weeks 3, 6, and 12
  Change from baseline of AUC 3-hr PPG
BMI | Week 12
  Change in Body Mass Index (BMI) from baseline
Lipids | Weeks 3, 6, and 12
  Change in serum lipid levels from baseline
Blood Pressure | Week 12
  Change in systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean arterial blood pressure (MAP) from baseline
hsCRP concentration | Weeks 3, 6, and 12
  Change in serum highly sensitive C-reactive protein (hsCRP) levels from baseline
C-peptide/insulin concentration | Weeks 3, 6, and 12
  Change in serum C-peptide or insulin levels from baseline
Fasting blood glucose concentration | Weeks 3, 6, and 12
  Change in fasting blood glucose from baseline
CGMS | Three days starting at Baseline, Weeks 3, 6, and 11
  Change in the AUC in Continuous Glucose Monitoring System (CGMS) from baseline
Change in oral hypoglycemic medication | Weeks 3, 6, and 12
  Change in oral hypoglycemic medication dosage

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Coastal Metabolic Research Center, Inc., Ventura, California
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Advanced Research Institute, Ogden, Utah